| Version 12 December 2023 |
|---|
| Pilot: Digital Therapeutic vs Education for the Management of Problematic Substance Use |
| NCT04974645 |

Descriptive statistics (means/standard deviations and frequencies/percentages) will be run to describe the sample demographics, clinical, substance use, and wellness outcomes, and programmatic feasibility, acceptability, and satisfaction; the balance achieved by randomization; and to determine the feasibility of including the Mini-International Neuropsychiatric Interview (MINI) to assess participants for a substance use diagnosis and phosphatidylethanol (PEth) as a biomarker indication of alcohol exposure during the 2-4 weeks prior to specimen collection in the RCT.